CLINICAL TRIAL: NCT03952325
Title: A Multicenter, Phase 2 Study of Tesetaxel Plus Three Different PD-(L)1 Inhibitors in Patients With Triple-Negative, Locally Advanced or Metastatic Breast Cancer and Tesetaxel Monotherapy in Elderly and Non-Elderly Adult Patients With HER2-Negative, Locally Advanced or Metastatic Breast Cancer
Brief Title: Tesetaxel Plus 3 Different PD-(L)1 Inhibitors in Patients With Triple-Negative MBC and Tesetaxel Monotherapy in Patients With HER2-Negative MBC
Acronym: CONTESSA TRIO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor has discontinued the development of tesetaxel
Sponsor: Odonate Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ODO-TE-B202
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: Tesetaxel; PD-(L)1 inhibitor; Triple-negative breast cancer; Locally advanced or metastatic breast cancer; Taxane; Metastatic breast cancer; Breast cancer; Combination of tesetaxel and PD-(L)1 inhibitors; HER2 negative; Oral chemotherapy; Central nervous system (CNS) metastases
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — tesetaxel; Nivolumab; pembrolizumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1, Arm A: Tesetaxel plus nivolumab (Experimental)
  Interventions: Drug: Tesetaxel; Drug: Nivolumab
- Cohort 1, Arm B: Tesetaxel plus pembrolizumab (Experimental)
  Interventions: Drug: Tesetaxel; Drug: Pembrolizumab
- Cohort 1, Arm C: Tesetaxel plus atezolizumab (Experimental)
  Interventions: Drug: Tesetaxel; Drug: Atezolizumab
- Cohort 2: Tesetaxel (Experimental)
  Interventions: Drug: Tesetaxel
- Cohort 3: Tesetaxel (Experimental)
  Interventions: Drug: Tesetaxel

INTERVENTIONS:
Drug: Tesetaxel — Tesetaxel at 27 mg/m2 orally Q3W
  Arms: Cohort 1, Arm A: Tesetaxel plus nivolumab
Drug: Tesetaxel — Tesetaxel at 27 mg/m2 orally Q3W
  Arms: Cohort 1, Arm B: Tesetaxel plus pembrolizumab
Drug: Tesetaxel — Tesetaxel at 27 mg/m2 orally Q3W
  Arms: Cohort 1, Arm C: Tesetaxel plus atezolizumab
Drug: Nivolumab — Nivolumab at 360 mg by intravenous infusion Q3W
  Arms: Cohort 1, Arm A: Tesetaxel plus nivolumab
Drug: Pembrolizumab — Pembrolizumab at 200 mg by intravenous infusion Q3W
  Arms: Cohort 1, Arm B: Tesetaxel plus pembrolizumab
Drug: Atezolizumab — Atezolizumab at 1,200 mg by intravenous infusion Q3W
  Arms: Cohort 1, Arm C: Tesetaxel plus atezolizumab
Drug: Tesetaxel — Tesetaxel at 27 mg/m2 orally Q3W
  Arms: Cohort 2: Tesetaxel; Cohort 3: Tesetaxel

SUMMARY:
CONTESSA TRIO is a multi-cohort, multicenter, Phase 2 study of tesetaxel, an investigational, orally administered taxane, in patients with metastatic breast cancer (MBC). In Cohort 1, approximately 200 patients with triple-negative MBC who have not received prior chemotherapy for advanced disease will be randomized 1:1:1 to receive tesetaxel plus either: (1) nivolumab; (2) pembrolizumab; or (3) atezolizumab. The primary efficacy endpoints for Cohort 1 are objective response rate (ORR) and progression free survival (PFS) in patients with programmed death-ligand 1 (PD-L1) positive status. In Cohort 2, approximately 60 elderly patients with human epidermal growth factor receptor 2 (HER2) negative MBC who have not received prior chemotherapy for advanced disease will receive tesetaxel monotherapy. The primary efficacy endpoints for Cohort 2 are ORR and PFS in patients with hormone receptor (HR)-positive, HER2-negative disease. In Cohort 3, approximately 60 non-elderly adult patients with HER2-negative MBC who have not received prior chemotherapy for advanced disease will receive tesetaxel monotherapy. The primary efficacy endpoints for Cohort 3 are ORR and PFS in patients with HR positive, HER2-negative disease.

DETAILED DESCRIPTION:
CONTESSA TRIO is a multi-cohort, multicenter, Phase 2 study of tesetaxel, an investigational, orally administered taxane, in patients with MBC.

Cohort 1:

Approximately 200 patients with triple-negative MBC who have not received prior chemotherapy for advanced disease will be randomized 1:1:1 to receive tesetaxel dosed orally at 27 mg/m2 once every three weeks (Q3W) plus either:

* Nivolumab at 360 mg by intravenous infusion Q3W;
* Pembrolizumab at 200 mg by intravenous infusion Q3W; or
* Atezolizumab at 1,200 mg by intravenous infusion Q3W.

Nivolumab and pembrolizumab (programmed cell death protein 1 [PD-1] inhibitors) and atezolizumab (a programmed death-ligand 1 [PD-L1] inhibitor) are immuno-oncology (IO) agents approved for the treatment of multiple types of cancer. Two of these agents, atezolizumab and pembrolizumab, have been approved by the U.S. Food and Drug Administration (FDA) as a first-line treatment for patients with triple-negative MBC. The primary efficacy endpoints for Cohort 1 are ORR and PFS in patients with PD-L1 positive status. The secondary efficacy endpoints are ORR and PFS in all patients, duration of response (DoR) and overall survival (OS).

Cohort 2:

Approximately 60 elderly patients with HER2-negative MBC who have not received prior chemotherapy for advanced disease will receive tesetaxel monotherapy dosed orally at 27 mg/m2 Q3W. The primary efficacy endpoints for Cohort 2 are ORR and PFS in patients with HR-positive, HER2-negative disease. The secondary efficacy endpoints are ORR and PFS in patients with triple-negative disease, DoR and OS.

Cohort 3:

Approximately 60 non-elderly adult patients with HER2-negative MBC who have not received prior chemotherapy for advanced disease will receive tesetaxel monotherapy dosed orally at 27 mg/m2 Q3W. The primary efficacy endpoints for Cohort 3 are ORR and PFS in patients with HR positive, HER2-negative disease. The secondary efficacy endpoints are ORR and PFS in patients with triple negative disease, DoR and OS.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients aged:

  * Cohort 1: ≥ 18 years old
  * Cohort 2: ≥ 65 years old
  * Cohort 3: ≥ 18 to < 65 years old
* Histologically or cytologically confirmed breast cancer
* Most recent biopsy must be HER2-negative
* Cohort 1 only: Most recent biopsy must be hormone receptor (HR) (estrogen receptor and progesterone receptor) negative
* Measurable disease per RECIST 1.1.

  * Patients with bone-only metastatic cancer must have a measurable lytic or mixed lytic-blastic lesion
  * Known metastases to the CNS are permitted but not required
* Documented (including de novo): (a) locally advanced breast cancer that is not considered curable by surgery and/or radiation; or (b) metastatic breast cancer
* Disease-free interval of at least 12 months after the completion of systemic neoadjuvant or adjuvant chemotherapy for patients previously treated with systemic chemotherapy for a tumor surgically resected with curative intent
* Cohorts 2 and 3 only: Prior endocrine therapy with or without a cyclin-dependent kinase (CDK) 4/6 inhibitor unless endocrine therapy is not indicated. Any prior targeted therapies are permitted. There is no limit to the number of prior endocrine therapies.
* Cohort 1 only: At Screening, patients must have documented evidence of positive PD-L1 expression as assessed via immunohistochemistry (IHC) scoring by local, regional, or central laboratory testing
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Adequate bone marrow, hepatic and renal function

Exclusion Criteria:

* Prior chemotherapy for locally advanced or metastatic disease
* Cohort 1 only: prior treatment with pembrolizumab, nivolumab, atezolizumab, any other PD-(L)1/PD-L2 inhibitor or a cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitor
* Current evidence or history of leptomeningeal disease
* Known human immunodeficiency virus infection, unless well controlled
* Known active hepatitis B or known active hepatitis C infection
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with Study participation or investigational product administration or may interfere with the interpretation of Study results
* Presence of neuropathy Grade > 1
* History of hypersensitivity to any of the Study drugs or any of their ingredients, as applicable
* Cohort 1 only:

  * Chronic autoimmune disease
  * Evidence of active, non-infectious pneumonia (eg, pneumonia due to autoimmune or connective tissue disease)
  * Treatment with a live vaccine within 30 days prior to the first dose of nivolumab, pembrolizumab or atezolizumab
  * History of active tuberculosis
  * Prior organ transplantation including allogeneic stem cell transplantation
  * Active infection requiring systemic therapy
  * Current or prior use of immunosuppressive medication within 7 days prior to Cycle 1, Day 1
  * Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
* Anticancer treatment, including endocrine therapy, radiotherapy (except stereotactic brain radiosurgery), chemotherapy or biologic therapy, ≤ 14 days prior to Enrollment
* Major surgery ≤ 28 days prior to Enrollment
* Less than 2 weeks or 5 plasma half-lives (whichever is greater) since last use of a medication or ingestion of an agent, beverage or food that is a known clinically relevant strong inhibitor or known clinically relevant inducer of the cytochrome P450 (CYP) 3A pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Cohort 1: ORR in patients with PD-L1 positive status | Approximately 2.0-3.0 years
Cohort 1: PFS in patients with PD-L1 positive status | Approximately 2.5-3.5 years
Cohort 2: ORR in patients with HR-positive, HER2-negative disease | Approximately 2.0-3.0 years
Cohort 2: PFS in patients with HR-positive, HER2-negative disease | Approximately 2.0-3.0 years
Cohort 3: ORR in patients with HR-positive, HER2-negative disease | Approximately 2.0-3.0 years
Cohort 3: PFS in patients with HR-positive, HER2-negative disease | Approximately 2.0-3.0 years

SECONDARY OUTCOMES:
Cohort 1: ORR in all patients | Approximately 2.0-3.0 years
Cohort 1: PFS in all patients | Approximately 2.0-3.0 years
Cohort 1: DoR | Approximately 2.5-3.5 years
Cohort 1: OS | Approximately 4.0-5.0 years
Cohort 2: ORR in patients with triple-negative disease | Approximately 2.0-3.0 years
Cohort 2: PFS in patients with triple-negative disease | Approximately 2.5-3.5 years
Cohort 2: DoR | Approximately 2.5-3.5 years
Cohort 2: OS | Approximately 4.0-5.0 years
Cohort 3: ORR in patients with triple-negative disease | Approximately 1.0-2.0 years
Cohort 3: PFS in patients with triple-negative disease | Approximately 1.5-2.5 years
Cohort 3: DoR | Approximately 2.5-3.5 years
Cohort 3: OS | Approximately 4.0-5.0 years

OTHER OUTCOMES:
Cohort 1: ORR by level of PD-L1 expression as determined by central PD-L1 testing | Approximately 2.0-3.0 years
Cohort 1: PFS by level of PD-L1 expression as determined by central PD-L1 testing | Approximately 2.5-3.5 years
Cohort 1: Central nervous system (CNS) ORR in patients with CNS metastases at baseline | Approximately 2.0-3.0 years
Cohort 1: CNS DoR in patients with CNS metastases at baseline | Approximately 2.5-3.5 years
Cohort 2: CNS ORR in patients with CNS metastases at baseline | Approximately 2.0-3.0 years
Cohort 2: CNS DoR in patients with CNS metastases at baseline | Approximately 2.5-3.5 years
Cohort 3: CNS ORR in patients with CNS metastases at baseline | Approximately 1.0-2.0 years
Cohort 3: CNS DoR in patients with CNS metastases at baseline | Approximately 1.5-2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph O'Connell, M.D., Study Director — Odonate Therapeutics, Inc.
Locations (12):
- United States (9):
  - Sarah Cannon Research Institute - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists and Research Institute, St. Petersburg, Florida
  - Florida Cancer Specialists and Research Institute - Panhandle Region, Tallahassee, Florida
  - Florida Cancer Specialists and Research Institute, West Palm Beach, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - New York Cancer and Blood Specialists, East Setauket, New York
  - West Cancer Center, Germantown, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
- Singapore (2):
  - John Hopkins Singapore International Medical Centre, Singapore
  - National Cancer Centre Singapore, Singapore
- Asan Medical Center, Seoul, South Korea